CLINICAL TRIAL: NCT02122354
Title: Data Collection and Analysis on Simulator Sickness Case Parameters in Susceptible Videogame Players
Brief Title: Triggers and Responses to Simulator Sickness in Videogame Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Marientina Gotsis, Research Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP-14-00222
Record Dates: First submitted 2014-04-17; First posted 2014-04-24 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Simulator Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Survey + videogame (Experimental): "Hide and Seek" videogame
  Interventions: Behavioral: "Hide and Seek" videogame

INTERVENTIONS:
Behavioral: "Hide and Seek" videogame

SUMMARY:
The objective of this research is the accumulation of gameplay data and simulator sickness background surveys for trend analysis, and individual simulator sickness trigger factor analysis for the test subjects involved. Rather than isolating specific variables for hypothesis formulation, this study will be attempting to collect an array of data that is a) both qualitative and quantitative, and b) observational and test subject-reported. The final results will consist of a list of possible trigger factors to avoid for individual subjects, and metrics showing the directional tendencies of players depending on the severity of their symptoms at the time.

The overall goal of this research is to better understand factors that contribute to simulator sickness, both in who it affects and why some gameplay experiences may cause it more than others. Operating from the basic assumption that the way a player moves through an environment affects how quickly that player gets sick, we will primarily be gathering data on how the player moves through the digital space and whether that behavior changes once they begin to feel sick.

ELIGIBILITY:
Inclusion Criteria:

* Survey participants should have some experience with playing videogames or similar interactive simulations on 2D displays.
* At least one-half of research participants should have experienced simulator sickness at some point in recent memory (within the past year) in response to a simulated experience.

Exclusion Criteria:

* Players under 18 will be excluded from participating in the experimental portion of the project.
* manual dexterity deficit or inability to use the gameplay interface
* Non-English speakers
* Acute state of illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Survey of triggers to simulator sickness in videogame players (global) | Baseline
  One-time questionnaire collecting demographic data, types of games participants play and any symptoms game players may have experienced in the past from up to 100 participants. This is a multiple choice tool created by the investigator.

SECONDARY OUTCOMES:
Survey of responses to simulator sickness in videogame players (global) | Baseline
  One-time questionnaire self-reported responses to simulator sickness for up to 100 participants. This is a multiple choice tool created by the investigator.
Real-time player responses to simulator sickness | During intervention
  Automated real-time in-game behavior data collection of up to to 30 minutes of game play. Specifically, directional movement up until simulator sickness onset, changes in movement behavior before and after sickness onset, first symptoms and time until onset. 10 participants will be selected for exposure to the intervention post-enrollment.

OTHER OUTCOMES:
Post-play simulator sickness rating | Post-exposure to intervention
  This is a questionnaire created by the investigator to rate simulator sickness induced by the intervention, compare it to other instances of simulator sickness and enumerate symptoms. Administered immediately after play.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lin, MFA, Principal Investigator — University of Southern California; Marientina Gotsis, MFA, Study Chair — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States